CLINICAL TRIAL: NCT04885127
Title: The Feasibility of Telehealth-Based Palliative Care Intervention and Digital Symptom Monitoring on Patients With AML Receiving Low-Intensity Induction Therapy
Brief Title: Feasibility of Telehealth Palliative Care and Digital Symptom Monitoring for Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Kavitha Ramchandran, Clinical Professor, Medicine - Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-60285; NCI-2022-03013 (Registry Identifier: CTRP)
Record Dates: First submitted 2021-05-01; First posted 2021-05-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Palliative Care
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): All patients enrolled in this trial will be referred to palliative care for planned monthly virtual visits, be instructed on the use of a digital application Noona that can be downloaded on their personal electronic device, and will be prompted to fill out symptom questionnaires using Noona prior to palliative care visits (required) as well as weekly (optional).
  Interventions: Other: Palliative Care + Digital Symptom Monitoring

INTERVENTIONS:
Other: Palliative Care + Digital Symptom Monitoring — Previously described in Arm description

SUMMARY:
AML is the most common leukemia diagnosed in adults. In spite of recent low-intensity therapies that have improved outcomes for older AML patients, AML remains associated with poor prognosis as well as high symptom burden. While the benefits of early palliative care as well as electronic PROs have been well-described in the oncology population, neither have been well-studied in the AML population, and have never been studied in combination. We propose a prospective, single-center, single-arm trial to evaluate the feasibility of a virtually-mediated supportive care model utilizing both electronic PROs and palliative care for patients with AML being treated with low-intensity therapy.

AIM1: is to evaluate and describe the feasibility of implementing early specialty palliative care referrals carried out via telehealth/video-based modalities in combination with digital symptom monitoring for patients recently diagnosed with acute myeloid leukemia (AML) and starting low intensity induction therapy.

AIM2: study the differences in health-related quality-of-life (HRQoL) metrics using patient-reported outcomes (PROs) in patients recently diagnosed with AML and starting low intensity induction therapy who receive early referral to telehealth/video-based palliative care visits compared to standard care.

AIM3: to explore the patient experience of patients with AML on low-intensity therapy, capture rates of advance care planning, hospice utilization, and hospital utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated for a diagnosis of acute myeloid leukemia at Stanford Cancer Center
* Patients determined to be candidates for low intensity induction therapy (not requiring hospitalization to administer treatment) by their leukemia physician
* Estimated life expectancy of 6 months
* Functional status at the level of at least being capable of limited self-care, confined to chair or bed for half the day or better
* Access to smartphone, tablet, or computer with capability to utilize a symptom tracking application

Exclusion Criteria:

* Relapsed or refractory AML
* Patients who have established care with palliative care previously
* Non-English-speaking, as the Noona application is developed in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of completed palliative care referrals and monthly visits | Through study completion, an average of 6 months
  This will be measured as a percentage of patients who overall complete the initial palliative care referral and at least 50% of their scheduled monthly visits
Rate of usage of digital symptom monitoring application, Noona | Through study completion, an average of 6 months
  This will be measured by the percentage of patients who complete at least 50% of Noona surveys associated with their palliative care visits

SECONDARY OUTCOMES:
Mean change in Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu) scores | Baseline, 3 months, and 6 months
  Health-related quality of life instrument used in patients with acute myeloid leukemia, minimum score 0, maximum score 176, higher scores indicating worse quality of life
Mean change in Hospital Anxiety and Depression Scale (HADS) scores | Baseline, 3 months, and 6 months
  Hospital Anxiety and Depression survey used to measure anxiety and depression, minimum score 0, maximum score 42, with higher scores indicating increased anxiety/depression
Mean change in Patient Health Questionnaire (PHQ)-9 scores | Baseline, 3 months, and 6 months
  Minimum score 0, maximum score 27, with higher scores indicating worse mood
Mean change in Satisfaction with Decision-Making Scale scores | Baseline, 3 months, and 6 months
  Minimum score 6, maximum score 25, with higher scores indicating improved satisfaction
Overall satisfaction with usage of Noona questionnaire | Baseline, 6 months
  Measured qualitatively, by whether patients strongly agree, somewhat agree, are neutral, somewhat disagree, or strongly disagree with statements regarding the Noona instrument

CONTACTS AND LOCATIONS:
Overall Officials: Kavitha Ramchandran, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No